CLINICAL TRIAL: NCT07218536
Title: The Burden of Atypical Hemolytic Uremic Syndrome and The Clinical Characteristics of Patients in Egyptian Hospitals A Multicenter, Observational, Retrospective Cohort Study in Egypt
Acronym: REACH
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D928BR00001
Record Dates: First submitted 2025-10-01; First posted 2025-10-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Atypical Hemolytic Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atypical hemolytic uremic syndrome (aHUS) is a rare, progressive, and life-threatening disease that occurs at any age, with incidence rate of 0.75 to 2.0 cases per million population per year. aHUS is a thrombotic microangiopathy (TMA) commonly caused by dysregulation of the complement system, affecting several organs, especially the kidneys. aHUS can be familial or sporadic, and approximately 50% to 60% of patients have specific identifiable genetic complement mutations and antibodies.

Although aHUS is a rare disease, it has a significant impact on the quality of life because of its poor prognosis: a 25% global mortality rate; more than 50% of untreated patients advance to endstage renal disease (ESRD); and more than 75% of adults with renal failure require prompt dialysis. The risk of relapse is also high in many patients, either in the native or transplanted kidneys, so long-term management and close monitoring are essential.

Advancements in aHUS therapies, especially the availability of anti-complement therapy, have enhanced the natural course of aHUS through hematologic remission induction, kidney function stabilization or improvement, and graft failure prevention. Since complement inhibitors are still unavailable in Egypt, it is important to understand the aHUS manifestations of pediatrics and adults in Egyptian hospitals, aiming for early diagnosis and proper management.

In this study, we primarily aim to describe the aHUS burden on the patients by gathering their demographic and clinical characteristics, documented disease course, and long-term complications. Our secondary objectives include an estimate of the prevalence of patients diagnosed with aHUS out of all patients with TMA and gathering information about the clinical outcomes of available therapies in real-world settings, as there is no data from the country on aHUS management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged one month or older who have been diagnosed with TMA between 01-Jan-2010 and 31-Dec-2023.

Exclusion Criteria:

* None. All records of patients with TMA will be screened for aHUS diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with TMA between 01-Jan-2010 and 31-Dec-2023 regardless of administered treatment. Medical records of all patients fulfilling the eligibility criteria will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical characteristics of patients with aHUS. | 10 Years
  Duration between the first aHUS treatment initiation and aHUS diagnosis

SECONDARY OUTCOMES:
The prevalence of patients diagnosed with aHUS | 10 Years
  The prevalence of patients diagnosed with aHUS among the total number of patients with TMA in the participating hospitals.
clinical outcomes of current treatment | 10 Years
  Overall survival rate (OS)
aHUS Treatment Patterns | 10 Years
  Treatment regimen(s)
aHUS Treatment Outcomes | 10 Years
  Overall Survival: defined as the proportion of people still alive at a given time point after treatment initiation

CONTACTS AND LOCATIONS:
Locations (7):
- Egypt (7):
  - Research Site, Al Mansurah
  - Research Site, Alexandria
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, New Cairo
  - Research Site, Tanta
  - Research Site, Zagazig

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/